CLINICAL TRIAL: NCT02557334
Title: Effects of Freeze Dried Strawberry Powder Supplementation on Vascular Function and Blood Markers of Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PKE STRAW II
Record Dates: First submitted 2015-09-18; First posted 2015-09-23 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: Strawberry Powder; Cardiovascular Disease Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose Strawberry Powder (Experimental): 40 g composed of 13 g freeze dried strawberry powder + 27 g placebo powder
  Interventions: Dietary Supplement: Low Dose Strawberry Powder
- High Dose Strawberry Powder (Experimental): 40 g freeze dried strawberry powder
  Interventions: Dietary Supplement: High Dose Strawberry Powder
- Placebo Powder (Placebo Comparator): 40 g color and taste matched placebo powder
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Low Dose Strawberry Powder — 40 g composed of 13 g freeze dried strawberry powder + 27 g placebo powder
  Arms: Low Dose Strawberry Powder
Dietary Supplement: High Dose Strawberry Powder — 40 g freeze dried strawberry powder
  Arms: High Dose Strawberry Powder
Dietary Supplement: Placebo Powder — 40 g color and taste matched placebo powder
  Arms: Placebo Powder

SUMMARY:
The purpose of this study is to evaluate the effects of freeze dried strawberry powder on LDL cholesterol, central and peripheral blood pressure, indices of arterial stiffness, and other lipid and lipoprotein concentrations. The investigators hypothesize that the bioactive compounds in freeze dried strawberry powder may elicit beneficial effects on LDL cholesterol, as well as blood pressure and arterial health.

DETAILED DESCRIPTION:
The proposed study design is a 3-period randomized crossover dose-response study to evaluate the effect of freeze dried strawberry powder supplementation on LDL-C and vascular health. Research participants will be overweight or obese (BMI 25-39 kg/m^2) but otherwise healthy adults with moderately elevated LDL-C (>116 mg/dL or >3.0mmol/L), blood pressure <160/100 mmHg, total cholesterol below 273 mg/dL for men and below 284 mg/dL for women, and triglycerides below 350 mg/dL. Subjects will be randomly assigned to three supplementation periods: 1) low dose freeze dried strawberry powder (13 g/d); 2) high dose freeze dried strawberry powder (40 g/d); and 3) a placebo powder. Each powder will be provided for 4-6 weeks, separated by a 2-week washout period between treatment periods. Baseline and endpoint testing will include blood collection and vascular testing.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 35-65 years of age
2. BMI ≥ 25 and ≤ 39 kg/m^2
3. LDL-C > 116 mg/dL
4. Total Cholesterol below 273 mg/dL for men and below 284 mg/dL for women
5. Triglycerides below 350 mg/d
6. Non-smokers
7. Blood pressure < 160/100 mmHg

Exclusion Criteria:

1. History of acute or chronic inflammatory conditions or heart disease, kidney disease, liver disease, autoimmune disorders, or thyroid disease (unless controlled by medication and blood results within the previous 6 months are provided)
2. History of diabetes mellitus (and/or a fasting glucose > 126 mg/dL at screening)
3. Stage II hypertension (blood pressure ≥ 160/100 mmHg)
4. Lactation, pregnancy, or desire to become pregnant during the study
5. Unwillingness to discontinue nutritional supplements, herbs, or vitamins, unless approved by investigator
6. Use of medications/supplements for elevated lipids, blood pressure, or glucose
7. Chronic use of non-steroidal anti-inflammatory or immunosuppressant medication
8. Conditions requiring the use of steroids
9. Unwillingness to refrain from blood donation prior to and during the study
10. Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator
11. Allergy or sensitivity to strawberries or any ingredient in the study powders

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
LDL-C | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  LDL-C values calculated using the Friedewald equation

SECONDARY OUTCOMES:
Central Blood Pressure | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Aortic (central) blood pressure measured using the SphygmoCor System
Peripheral Blood Pressure | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Peripheral blood pressure measured using the SphygmoCor System
Augmentation Index | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Augmentation index measured using the SphygmoCor System
Pulse Wave Velocity | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Pulse wave velocity measured using the SphygmoCor System
Total Cholesterol | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Total cholesterol values determined by enzymatic procedures
Triglycerides | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Triglyceride values determined using enzymatic procedures
HDL-C | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  HDL-C will be estimated according to the modified heparin-manganese procedure
Oxidized LDL (oxLDL) | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  Plasma concentrations of oxLDL will be measured using ELISA kits
Malondialdehyde (MDA) | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  MDA will be measured using the thiobarbituric acid reactive substances (TBARS) assay
High Sensitivity C Reactive Protein (hs-CRP) | Change from baseline after 4 week treatments of low dose, high dose, and placebo strawberry beverage
  hs-CRP will be measured by latex-enhanced immunonephelometry

CONTACTS AND LOCATIONS:
Overall Officials: Penny Kris-Etherton, PhD, RD, Principal Investigator — Penn State University
Locations (1):
- Penn State CRC, University Park, Pennsylvania, United States